

# Safety and Effectiveness of Edwards Lifesciences SAPIEN 3 Transcatheter Heart Valve (THV) in the Chinese Population

NCT03466918

June 22, 2017

# Table of Contents

| 1. | Information of sponsors | 5 |
|---|---|---|
| | 1.1 Name of sponsors: | 5 |
| | 1.2 Address of sponsors: | 5 |
| | 1.3 Contact information of sponsors: | 5 |
| | 1.4 Relevant qualification documents of sponsors: | 5 |
| | 1.5 Name, address, contact information, and relevant qualification documents of agents: | 5 |
| 2. | List of all clinical trial institutions and investigators for multicenter clinical trials | 5 |
| 3. | Purpose and contents of clinical trials | 6 |
| | 3.1 Purpose | 6 |
| | 3.2 Contents | 6 |
| 4. | Background information of clinical trials | 7 |
| | Disease Process | 7 |
| | Alternative Therapies/Techniques. | 8 |
| | Transcatheter Aortic Valve Implantation (TAVI) | 8 |
| 5. | Characteristics, structure and composition, operating principle, mechanism of action, and tes | st range |
| of p | product | 8 |
| | 5.1 Product characteristics | 9 |
| | SAPIEN 3 Transcatheter Heart Valve | 9 |
| | 5.2 Structure and composition, operating principle, mechanism of action of product | 9 |
| | Commander Delivery System | 10 |
| | Expandable Introducer Sheath Set | 10 |
| | Edwards Transfemoral Balloon Catheter | 10 |
| | Loader | 10 |
| | Crimper | 10 |
| | Qualcrimp | 10 |
| | 5.3 Trial range | 11 |
| 6. | Indications of products and contraindications, and matters needing attention | 11 |
| 7. | Overall design | 11 |
| | 7.1 Trial design | 11 |
| | 7.1.1 Trial purpose | 11 |
| | 7.1.2 Selection of test methods and reasons | 12 |
| | 7.1.3 Measures for reducing and avoiding bias | 12 |
| | 7.1.4 Selection of subjects (including selection of control group if necessary) | 12 |
| | 7.1.5 Patient Screening and Data Collection | 14 |
| | Screening | 17 |
| | Baseline | 17 |
| | Procedure | 18 |
| | Post-Procedure | 20 |
| | Discharge Visit | 20 |
| | Follow-Up Visits | 21 |
| | 30-Day Visit | 22 |
| | 6 Month Visit | 22 |
| | 1 Year Visit | 22 |

| | 2-5 Ye | ear Annual Follow-up Visit | 23 |
|---|---|---|---|
| | Misse | d Visits | 23 |
| | Stand | ard of Care | 23 |
| | 7.1.6 | Safety and Effectiveness evaluation methods | 24 |
| | 7.2 | Test process | 25 |
| | 7.2.1 | Test flowchart | 25 |
| | 7.2.2 | Specification for use of devices | 25 |
| | Study | Device | 26 |
| | Storag | ge & Labeling | 26 |
| | Devic | e Accountability | 26 |
| | 7.3 | Monitoring Plan | 26 |
| 8. | Sta | tistical considerations | 27 |
| | 8.1 | Statistical design, method, and analysis procedures | 27 |
| | 8.2 | Sample Size | 27 |
| | 8.3 | Expected expulsion rate | 28 |
| | 8.4 | Statistical method for all data, together with deficient, unused or fault data (including of | drop out |
| | and w | ithdrawal) and method for treating unreasonable data | • |
| | 8.5 | Procedures for reporting deviation from the original statistical plan | |
| | 8.6 | Criteria and reasons for selection of subjects incorporated into analysis | 28 |
| 9. | Da | a Management | |
| | 9.1 | Data Collection | 29 |
| | 9.2 | Missing Data | 29 |
| 10. | Fea | sibility Analysis | 29 |
| | 10.1 | Successful possibility analysis | 29 |
| | 10.2 | Analysis of the possibility of failure | 30 |
| 11. | Qu | ality control of clinical trials | 30 |
| 12. | Eth | ical issues and informed consent for clinical trials | 30 |
| | 12.1 | Ethical considerations | 30 |
| | 12.2 | Examination and approval of clinical trial protocol | |
| | 12.3 | Informed consent process and text of informed consent | |
| 13. | Pro | visions on adverse event and device defect report | 31 |
| | 13.1 | Adverse events | |
| | 13.2 | Serious Adverse Events | 32 |
| | 13.3 | Reporting procedure and information of contact | 32 |
| | Sourc | e Documents | |
| | Invest | igator Assessment Responsibilities | 32 |
| | | or Assessment Responsibilities | |
| | Medic | eal Reviewer Responsibilities | 33 |
| | Devic | e Deficiency and Vigilance Reporting | 33 |
| 14. | | visions on deviation from clinical trial protocol and correction of clinical trial protocol | |
| 15. | | ect access to source data and files | |
| | Recor | ds | 34 |
| | Recor | d Retention Policy | 34 |
| 16. | Fin | ance and insurance | 34 |
| | Clinic | al Trial Funding | 34 |

| Clinical Trial Insurance | |
|---|---|
| 17. Contents to be covered by clinical trial reports | |
| 18. Principle of medical confidentiality | |
| 19. Provisions on publication of clinical trial results | |
| 20. Responsibilities of all parties | |
| General Study Organization | |
| Medical Reviewers | |
| Echocardiography Core Laboratory | |
| Clinical Sites | |
| Statement of Investigator | |
| Appendix A | Defnitions |
| Appendix B | |
| Appendix C | NIH Stroke Scale |
| Appendix D | Modified Rankin Score |
| Appendix E | Frailty Index |
| Appendix F | 6MWT |
| Appendix G | KCCQ |
| Appendix H | Clinical Trial Report Content |

# 1. Information of sponsors

# 1.1 Name of sponsors:

Edwards Lifesciences LLC

# 1.2 Address of sponsors:

One Edwards Way Irvine, CA 92614 USA

# 1.3 Contact information of sponsors:

One Edwards Way

Irvine, CA 92614 USA

# 1.4 Relevant qualification documents of sponsors:

Edwards Lifesciences LLC

ISO 13485:2003

Number: 3805474

# 1.5 Name, address, contact information, and relevant qualification documents of agents:

Edwards (Shanghai) Medical Products Co., Ltd

Email contacts:

Chinese Business Certificate No: 913100006074327581

# 2. List of all clinical trial institutions and investigators for multicenter clinical trials

| Study Consultant | Prof Runlin GAO |
|---|---|
| National Principal | Prof Junbo GE |
| Investigator | PTOI JUHOO GE |
| National Co-PI | Prof. Yuejin YANG Prof. Jianan WANG Prof. Mao CHEN |

| Code number of clinical trial institution | Name of clinical trial institution | Investigator | Technical<br>title | Contact |
|---|---|---|---|---|
| S-ZS | Zhongshan Hospital<br>Fudan University | Junbo GE | Professor | |
| S-FW | Fuwai Hospital,<br>CAMS&PUMC | Yongjian<br>WU | Professor | |

| S-ZJ | The Second Affiliated Hospital of Zhejiang University School of Medicine | Jianan<br>WANG | Professor |
|---|---|---|---|
| S-HX | WestChina Hospital,<br>Sichuan University | Mao CHEN | Professor |

#### 3. Purpose and contents of clinical trials

#### 3.1 Purpose

The purpose of this trial is to evaluate the safety and effectiveness of the SAPIEN 3 transcatheter heart valve implantation (TAVI) in Chinese patients with symptomatic severe calcific aortic stenosis who are considered at high risk for surgical valve replacement. Clinical data will be submitted for the purposes of obtaining Chinese regulatory approval.

#### 3.2 Contents

This is a prospective, single-arm, multi-center study to assess the safety and effectiveness of the SAPIEN 3 THV. A minimum of 50 patients (maximum of 60 patients) with symptomatic severe calcific aortic stenosis requiring transcatheter aortic valve implantation (TAVI), who are considered high risk for surgical valve replacement and who receive a SAPIEN 3 THV.

Study endpoints include:

#### **Primary Endpoint**

The primary endpoint is all-cause mortality at 30 days post-index procedure.

# Secondary Endpoints

#### Safety Endpoints

- Cardiovascular and non-cardiovascular mortality at 72 hours (peri-procedural) and 30 days
- Stroke at 30 days
- TIA at 30 days
- All-cause mortality & disabling stroke at 30 days
- Vascular complications (major) at 30 days
- Bleeding complications (life threatening or disabling, and major) at 30 days
- Myocardial infarction at 30 days
- Acute kidney injury at 30 days (stages II and III)
- Coronary obstruction requiring intervention at 30 days
- Arrhythmia and conduction disturbance at 30 days
- Permanent pacemaker implantation at 30 days
- Valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVR) at 30 days

- Mitral valve apparatus damage or dysfunction at 30 days
- Unplanned use of cardiopulmonary bypass (CPB) during TAVI implant procedure
- Pericardial tamponade at 30 days
- Endocarditis at 30 days
- Valve thrombosis at 30 days
- Valve malposition (migration, embolization, and ectopic deployment) at 30 days
- Ventricular septal perforation at 30 days

#### Device and Procedure Success Composite

- Absence of procedural mortality AND
- Correct positioning of a single prosthetic heart valve into the proper anatomic location AND
- Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20mmHg or peak velocity <3m/s, AND no moderate or severe prosthetic valve regurgitation) at 30 Days

# Efficacy

- New York Heart Association (NYHA) Classification at 30 days
- Hemodynamic valve performance evaluation by echocardiography for aortic valve stenosis and aortic valve regurgitation (paravalvular & central) at 30 Days as determined by Echo core lab

# Quality of Life

• KCCQ at 30 days

#### 4. Background information of clinical trials

Prolonged average life expectancy has resulted in an aging population and consequently, an increase in the number of patients with acquired, calcific, severe, symptomatic aortic stenosis (AS). The standard of care therapy for patients suffering from severe AS is aortic valve replacement surgery (AVR). In the aged population, many patients are too sick to be operated or have co-morbidities that preclude the option for surgery [1].

AS is a progressive, debilitating and life-threatening disease if left untreated. Affected individuals are typically > 65 years of age. The pathology involves progressive calcification of the leaflet bodies which limits normal cusp opening during systole. Cellular aging and degeneration have been implicated in this form of the disease and diabetes mellitus and hypercholesterolemia are risk factors.

#### **Disease Process**

The pathophysiology of AS includes an increase in afterload, progressive hypertrophy of the left ventricle, and a decrease in systemic and coronary blood flow as consequences of valve obstruction. Typically, patients with AS are free from cardiovascular symptoms (e.g. angina, syncope and/or heart failure) until late in the course of the disease. However, once symptoms manifest, the prognosis is poor, especially when associated with congestive heart failure.

Death in general, including sudden death, occurs primarily in symptomatic patients. Survival analyses have demonstrated that the interval from onset of symptoms to time of death is approximately two years in patients with heart failure, three years in those with syncope, and five years in those with angina [2]. Among symptomatic patients with moderate-to-severe AS treated medically, mortality rates after the onset of symptoms were approximately 25% at 1 year and 50% at 2 years and more than 50% of deaths were sudden [3].

Grading the severity of AS is based on a variety of hemodynamic and natural history data. According to the ACC/AHA guideline authors, AS is best described as a continuum. In patients with moderate-to-severe AS, valve area may decline up to 0.3 cm<sup>2</sup> per year and the systolic pressure gradient across the valve can increase by as much as 15-19 mmHg per year, with a higher rate of progression observed in elderly patients with coronary artery disease

(CAD) and chronic renal insufficiency [4]. Relief of aortic valve obstruction typically results in an improvement of symptoms, hemodynamic parameters, and global left ventricle systolic function, as well as reversal of left ventricular hypertrophy [4,5].

# Alternative Therapies/Techniques

Treatment options for patients suffering from symptomatic aortic stenosis, prior to the introduction of transcatheter aortic valve implant (TAVI), included palliation of symptoms without valve replacement (non-surgical standard therapy), or surgical aortic valve replacement (AVR). Treatment options were determined by patient risk for morbidity or mortality after surgery and patient choice. Non-surgical treatment options, including balloon aortic valvuloplasty, did not provide sustained hemodynamic improvement and have led to poor quality of life and shortened life expectancies [5-7]. Patients considered poor candidates for AVR typically present with significant multiple morbidities or anatomical limitations [8].

Patient frailty may also contribute to the decision to forego surgery. Surgical AVR has demonstrated excellent long term outcomes for patients with a ortic valve stenosis, even in high risk populations (STS PROM > 10) [5-7, 9-11].

# Transcatheter Aortic Valve Implantation (TAVI)

Transcatheter aortic valve implantation (TAVI) was first performed in man in 2002 [12], followed by clinical trials and approval for commercialization in Europe in 2007 [13, 14]. It is currently estimated that approximately 300,000 patients have undergone TAVI worldwide. The Edwards THV global clinical research program includes more than 30,000 patients enrolled in 18 clinical studies that include first-in-man, feasibility, and pivotal studies as well as randomized controlled trials and post market registries. Results and outcomes from these trials have been publically reported at medical congresses and in peer-reviewed scientific journals [15-22]. The randomized PARTNER I Trial produced the most conclusive evidence of safety and effectiveness of the Edwards SAPIEN THV in high surgical risk (Cohort A) and inoperable (Cohort B) patients with severe, symptomatic aortic stenosis [23,24]. The PARTNER II trial demonstrated safety and effectiveness of the second and third generation valves, the SAPIEN XT THV and SAPIEN 3, respectively, in intermediate risk, high risk and inoperable patients [25,26].

# 5. Characteristics, structure and composition, operating principle, mechanism of action, and test range of product

#### 5.1 Product characteristics

#### SAPIEN 3 Transcatheter Heart Valve

The Edwards SAPIEN 3 Transcatheter Heart Valve (Figure 1) is indicated for use in patients with severe, symptomatic, calcified aortic stenosis.

The Edwards SAPIEN 3 transcatheter heart valve (THV) is comprised of a balloon-expandable, radiopaque, cobalt-chromium alloy frame, trileaflet bovine pericardial tissue valve, and polyethylene terephthalate (PET) fabric skirt. It is treated according to the Edwards ThermaFix process, and is packaged and terminally sterilized in glutaraldehyde.

Figure 1. SAPIEN 3 Transcatheter Heart Valve (THV)



# 5.2 Structure and composition, operating principle, mechanism of action of product

The SAPIEN 3 THV is provided with the Commander Delivery System and other components. Table 1 summarises the components that may be provided in the kit.

Table 1. SAPIEN 3 THV Commander Kit

| Product Name | 20 mm System | 23 mm System | 26 mm System | 29 mm System |
|---|---|---|---|---|
| | | Model/REF | | |
| Kit | S3TF120 | S3TF123 | S3TF126 | S3TF129 |
| Edwards SAPIEN 3<br>Transcatheter Heart<br>Valve | 9600TFX20<br>(20 mm) | 9600TFX23<br>(23 mm) | 9600TFX26<br>(26 mm) | 9600TFX29<br>(29 mm) |
| Commander<br>Delivery System <sup>1</sup> | 9610TF20 | 9610TF23 | 9610TF26 | 9610TF29 |

| Edwards Expandable Introducer Sheath Set ("eSheath") | 9610ES14 | 9610ES14 | 9610ES14 | 9610ES16 |
|---|---|---|---|---|
| Edwards<br>Transfemoral<br>Balloon Catheter | 9350BC16 | 9350BC20 | 9350BC23 | 9350BC25 |
| Crimper | 9600CR | 9600CR | 9600CR | 9600CR |
| Inflation Devices (x2) | 96402 | 96402 | 96402 | 96406 |

<sup>&</sup>lt;sup>1</sup>Includes a Loader, Qualcrimp Crimping Accessory, and 2-piece Crimp Stopper

#### Commander Delivery System

The Edwards Commander Delivery System consists of a balloon catheter for deployment of the THV and a Flex Catheter to aid in valve alignment to the balloon, tracking and positioning of the THV. The delivery system includes a tapered tip to facilitate crossing of the aortic valve. The handle contains a FlexWheel to control flexing of the Flex Catheter, and a Balloon Lock and Fine Adjustment Wheel to facilitate valve alignment and positioning of the valve within the aortic annulus. A stylet is included within the guidewire lumen of the delivery system. The Balloon Catheter has radiopaque Valve Alignment Markers defining the working length of the balloon. A radiopaque Center Marker in the balloon is provided to help with valve positioning. A radiopaque Triple Marker proximal to the balloon indicates the Flex Catheter position during deployment.

#### Expandable Introducer Sheath Set

The Edwards eSheath Introducer Set is intended for introduction of interventional devices in the vascular system. The product is intended for use by physicians trained and experienced in interventional techniques. Standard techniques for placement of vascular access sheaths should be employed.

#### Edwards Transfemoral Balloon Catheter

The balloon catheter is indicated for dilation of stenotic native aortic valve leaflets.

#### Loader

The loader (packaged with the Edwards Commander delivery system) is used to aid insertion of the delivery system into the sheath, and may be removed to utilize the full working length of the inserted device

#### Crimper

The crimper reduces the diameter of the THV to mount it to the delivery system. The crimper is comprised of a compression mechanism that is closed with a handle located on the housing. The crimper is used with a 2-piece crimp stopper (packaged with the delivery system) to correctly crimp the THV.

#### Qualcrimp

The Qualcrimp crimping accessory (packaged with the Qualcrimp delivery system) is used during crimping of the THV.

#### Inflation Device

An inflation device with locking mechanism may be used during native valve predilation and THV deployment.

#### 5.3 Trial range

The THV is intended to be implanted in a native annulus size range comparable to the following measurements:

Table 1. SAPIEN 3 Annulus and Valve Sizing

| Native Valve | Native Valve Ar | nulus size (CT) | |
|---|---|---|---|
| Annulus Size (TEE) | Area | Area Derived<br>Diameter | THV size |
| 16-19 mm | 273-345 mm <sup>2</sup> | 18.6-21.0 mm | 20 mm |
| 18-22 mm | 338-430 mm <sup>2</sup> | 20.7-23.4 mm | 23 mm |
| 21-25 mm | 430-546 mm <sup>2</sup> | 23.4-26.4 mm | 26 mm |
| 24-28 mm | 540-683 mm <sup>2</sup> | 26.2-29.5 mm | 29 mm |

# 6. Indications of products and contraindications, and matters needing attention

These devices must always be used according to the current Instructions for Use (IFU) provided with each product

#### Indications

The Edwards SAPIEN 3 valve, Edwards Commander delivery system and accessories are indicated for use in patients with severe, symptomatic, calcific aortic valve stenosis who are considered at high risk for surgical valve replacement

#### Contraindications

Use of the Edwards SAPIEN 3 valve with the Edwards Commander delivery system and accessories is contraindicated in patients with:

- Evidence of intracardiac mass, thrombus, vegetation, active infection or endocarditis
- Inability to tolerate anticoagulation/antiplatelet therapy

#### 7. Overall design

# 7.1 Trial design

#### 7.1.1 Trial purpose

The purpose of this trial is to evaluate the safety and effectiveness of the SAPIEN 3 transcatheter heart valve implantation (TAVI) in Chinese patients with symptomatic severe calcific aortic stenosis who are considered at high risk for surgical valve replacement. Clinical data will be submitted for the purposes of obtaining Chinese regulatory approval.

#### 7.1.2 Selection of test methods and reasons

This is a prospective, single-arm, multi-center study to assess the safety and effectiveness of the SAPIEN 3 THV. Up to 60 patients will be enrolled and implanted with the device at four sites in China over an estimated six-month enrolment period with a follow-up period to 5 years. The study is expected to last 5.5 years.

An Echocardiography Core Lab will be established for standardizing echocardiographic secondary endpoints. A Medical Reviewer will review all endpoint-related adverse events.

#### 7.1.3 Measures for reducing and avoiding bias

An independent Echocardiography Core Lab will be established for standardizing echocardiographic secondary endpoints. A Medical Reviewer will review all endpoint-related adverse events independently.

#### 7.1.4 Selection of subjects (including selection of control group if necessary)

To ensure that a minimum of 50 patients are implanted with the SAPIEN 3 THV and complete the 30 Day follow-up for Primary Endpoint, up to 60 patients will be enrolled and implanted with SAPIEN 3 THV. Each site may not contribute more than 25 implanted patients to the study population. All patients will be followed for 5 years.

Enrolment will be closely monitored to ensure not more than 60 patients are implanted with SAPIEN 3 THV.

#### 7.1.4.1 Inclusion Criteria

Patients must meet all of the Inclusion Criteria in order to participate in the study

- Subjects who are considered to be operable and high risk for surgical valve replacement: STS Score ≥ 8 and ≤ 15 or Logistic EuroSCORE ≥ 15 and ≤ 40. If STS Score is below 8 and Logistic EuroSCORE is below 15, patients should have other clinical or anatomical risk factors that would be considered high risk for surgery and documented by the heart team
- 2. Severe symptomatic calcific aortic stenosis requiring aortic valve replacement characterized by one or more of the following within 60 days prior to the index procedure: AVA < 0.8 cm<sup>2</sup>, Indexed AVA <0.5 cm<sup>2</sup>/m<sup>2</sup>, mean gradient > 40mmHg, or peak aortic jet velocity > 4.0m/sec.
- 3. NYHA Functional Class II or greater.
- 4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the EC of the respective clinical site.
- 5. The study patient agrees to comply with all required post-procedure follow-up visits.
- 6. Native aortic valve annulus area between 273 mm<sup>2</sup> 683 mm<sup>2</sup> as measured by CT.
- 7. Native a ortic annulus diameter between 18.6 mm 29.5 mm as measured by CT.

# 7.1.4.2 Exclusion Criteria

Patients must not meet any of the Exclusion Criteria in order participate in the study

- Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [(defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
- 2. Aortic valve is a congenital unicuspid or is non-calcified.
- 3. Aortic valve is bicuspid and the patient is less than 60 years old, or the aortic valve is bicuspid with no raphe (Sievers classification type 0)
- 4. Anomalous coronary artery that would interfere with proper placement of the valve.
- 5. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
- 6. Pre-existing mechanical or bioprosthetic valve in any position.
- 7. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure. Implantation of a permanent pacemaker or ICD is not considered exclusion criteria.
- 8. Any patient with a balloon valvuloplasty (BAV) within 30 days of the procedure (unless BAV is a bridge to procedure after a qualifying echocardiogram).
- 9. Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mL).
- 10. Renal insufficiency (creatinine > 3.0 mg/dL) and/or renal replacement therapy at the time of screening.
- 11. Untreated clinically significant coronary artery disease requiring revascularization.
- 12. Emergency interventional/surgical procedures within one month (30 days) prior to the TAVI procedure.
- 13. Hypertrophic cardiomyopathy (HCM with myocardium more than 1.5cm without an identifiable cause) with or without obstruction (HOCM).
- 14. Severe ventricular dysfunction with LVEF < 20%.
- 15. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
- 16. Active upper GI bleeding within 3 months (90 days) prior to procedure.
- 17. A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
- 18. Stroke or transient ischemic attack (TIA) within 3 months (90 days) of the procedure.
- 19. Estimated life expectancy < 12 months (365 days) due to carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease.
- 20. Significant aortic disease, including marked tortuosity (hyperacute bend), aortic arch atheroma [especially if thick (> 5 mm), protruding or ulcerated] or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta.
- 21. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
- 22. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
- 23. Active bacterial endocarditis within 6 months (180 days) of procedure, with our without treatment.

#### 7.1.4.3 Standard and procedures for stopping tests/trial treatment

The Sponsor has the right to discontinue a site or terminate the trial for the following reasons:

- The Sponsor may terminate the study for safety reasons
- A decision on the part of the Sponsor to suspend or discontinue testing, evaluation, or development of the product for any reason
- The Sponsor may decide to close a study site when the Investigator fails to enroll patients during the enrolment period
- Failure of the Investigator to comply with pertinent regulations of appropriate regulatory authorities
- Insufficient adherence to protocol requirements
- Submission of knowingly false information from the research facility to the Sponsor, the Sponsor's representatives or appropriate regulatory authorities

If the study is terminated early, all specified follow-up data on subjects enrolled prior to termination will be collected and reported

# 7.1.4.4 Enrollment period and study duration

Up to 60 patients will be enrolled and implanted with the device at four sites in China over an estimated six month enrolment period with a follow-up period to 5 years. The study is expected to last 5.5 years

#### 7.1.5 Patient Screening and Data Collection

# 7.1.5.1 Patient Screening and Enrolment

The study site shall have a committed Heart Team involved in the screening process. The Heart Team will include at least two cardiac surgeon, one interventional cardiologist, one radiologist, and one anesthesiologist but could also include (without being limited to) the following specialties:

- Echocardiography
- Gerontology

The screening of patients in cardiovascular and cardiac surgery departments will be conducted by one or more delegated study team members. The study team will be responsible for ensuring and reporting study patient screening for study eligibility. Cumulative screening and enrollment logs will be maintained by study sites. Reasons for screen failures will be documented in study logs.

To accommodate the implant procedure learning curve, a roll-in strategy will be available. Each study site will be allowed up to two roll-in patients. Edwards Lifesciences will document if the patient is a roll-in patient before the implant procedure begins. Roll-in patients will complete all study visits and procedures, and not be counted toward the 60 implanted patients.

In addition, the Heart Team will be required to assess all patients for study inclusion to ensure compliance to surgical risk criteria, screening procedures to assess valve size and delivery method, and other inclusion/exclusion criteria. After heart team identifies a patient, the Sponsor will review and confirm eligibility during the case review process.

All patients who sign a study informed consent will be entered into the database. Subjects will be included

in analysis of the trial if an Edwards' investigational device is inserted into the patient. Only patients that leave the procedure room with a SAPIEN 3 THV in place will be counted toward the 60 implanted patients.

#### 7.1.5.2 Data Collection

Study subjects will undergo screening and pre-procedure visits, and then follow-up visits at Discharge, and 30 Days (+14 days) for Endpoint analysis. Long-term follow-up data is collected at 6 Months (+/- 30 days), 1 Year (+/- 60 days), 2 Years (+/- 60 days), 3 Years (+/- 60 days), 4 Years (+/- 60 days), and 5 Years (+/- 60 days).

The Study Visit Schedule is outlined in Table 4 for enrolled subjects for the duration of the study from Screening and Baseline through the 30 Day visit (Primary Endpoint) and 5 year follow-up visits.

Table 2. Study Visit Schedule

| | Screening | Baseline<br>(≤30 days of procedure) | Procedure | Post-Procedure (Within 48 hours) | Discharge | 30 Day Follow-Up<br>(+14 days) | 6 Month (+/-30<br>days) | 1 Year (+/-60 days) | 2-5 Years (+/-60 days) |
|---|---|---|---|---|---|---|---|---|---|
| <b>Informed Consent</b> | X | | | | | | | | |
| Medical History | X | | | | | | | | |
| Physical Exam | X | | | | X | X | | X | X |
| CSS Angina | X | | | | X | X | | X | X |
| NYHA<br>Classification | X | | | | X | X | | X | X |
| STS Risk Score, Logistic EuroSCORE, and EuroSCORE II | X | | | | | | | | |
| Operability Risk<br>Assessment | X | | | | | | | | |
| Cardiac<br>Medications | | X | X | X | X | X | X | X | X |
| Adverse Event Assessment <sup>1</sup> | | | X | X | X | X | X | X | X |
| Frailty Assessment | | X | | | | | | | |
| NIH Stroke Scale | | $X^2$ | | $X^2$ | $X^2$ | $X^2$ | | | |
| Modified Rankin<br>Scale | | $X^2$ | | $X^2$ | $X^2$ | $X^2$ | | | |
| Six Minute Walk<br>Test (6MWT) | | $X^3$ | | | | $X^3$ | | | |
| KCCQ<br>Questionnaire | | X | | | | X | | | |
| | | | | Labs | | | | | |

| Hemoglobin, Hematocrit, Platelet Count and White Blood Cells | | X | | X | X | X | | |
|---|---|---|---|---|---|---|---|---|
| PTT or PT/INR | | X | | X | X | | | |
| CK/CK-MB<br>and/or Troponins | | $X^4$ | | X <sup>5</sup> | | X | | |
| Creatinine | | X | | X | X | X | | |
| Liver Panel (ALT, AST) | | X | | | | | | |
| Albumin | | X | | | | X | | |
| | | | Non- | Invasive Te | sts | | | |
| ECG | | X | | X | X | X | X | |
| Chest X-ray | | X | | | | | | |
| Transthoracic | | | | | | | | |
| Echocardiogram | X | | | | X | X | X | X |
| (TTE) <sup>6</sup> | | | | | | | | |
| Fluoroscopic | | | | | | 7 | 7 | 7 |
| imaging implanted | | | X | | | $X^7$ | $X^7$ | $X^7$ |
| valve | | | Too | vasive Tests | | | | |
| CT | | | 111/ | vasive tests | | | | |
| Thoracic/Abdome n with visualization of iliac and femoral arteries | X | | | | | | | |
| Cardiac Catheterization or CT angiogram | X | | | | | | | |
| Supra-aortic Angiogram or (TEE) | X | | X | | | | | |
| Invasive<br>hemodynamics | | | X | | | | | |

<sup>&</sup>lt;sup>1</sup> Collection of adverse events begins when the patient starts the procedure. This is defined as when anesthesia is first administered <sup>2</sup>Every effort should be made to have a neurologist or neurology fellow perform the neurological assessments. If the neurologist or neurology fellow is not available, a certified team member may perform the tests.

<sup>&</sup>lt;sup>3</sup>Patients are exempt from the 6 Minute Walk Test if they are contraindicated to complete the test. Contraindications must be documented in medical notes.

 $<sup>^4</sup>$ Baseline CK/CKMB and/or Troponins are required  $\leq$  72 hours before the procedure.

<sup>&</sup>lt;sup>5</sup>Post Procedure CK/CKMB and/or Troponins are required at 3 different time intervals: 1) the first lab draw post procedure (within 8 hours of exiting the cath lab or operating room) 2) the second lab draw 6 – 8 hours after the first lab draw 3) the third lab draw 6 – 8 hours after the second lab draw.

#### Screening

The following screening data will be collected for all study patients to assess eligibility as per standard of care:

- Operability Risk Assessment
- Medical history, pertinent physical examination [include blood pressure, height, weight and all major systems findings]
- NYHA functional classification
- CSS Angina classification
- Risk assessment (STS Risk Score, Logistic EuroSCORE, and EuroSCORE II)
- Non-Invasive Studies (must be completed within 60 days before procedure date)
- Comprehensive transthoracic echocardiogram (TTE) (transesophageal echocardiogram (TEE) may be used as an alternative)

Invasive Studies (must be completed before the procedure date)

- Cardiac and abdominal CT angiogram of high quality with complete visualization to complete measurements of the aortic valve, aortic arch, both iliac and femoral arteries to the aorta. In the situation where patients have compromised renal function that precludes the use of contrast agents, MR imaging may be used as an alternative to CT (≤180 days before procedure)
- Left heart catheterization to assess the severity of aortic stenosis and severity of coronary artery disease (≤180 days before procedure)

If any assessments need to be completed or repeated outside of standard of care, a patient will need to sign a Patient Informed Consent prior to completing assessments.

#### **Baseline**

Assessments and laboratory tests are required to be completed within 30 days prior to the procedure date. Assessments and laboratory tests completed outside of the 30 days will need to be repeated. If completed outside of standard of care, then a Patient Informed Consent Form will need to be signed first.

The following Baseline data will be collected for all study patients prior to procedure:

- Current cardiac medications and all medications given for cardiovascular effect;
- Neurological assessment
  - o National Institutes of Health Stroke Scale (NIHSS) (Appendix C)
  - o Modified Rankin Scale (mRS) (Appendix D)
- Frailty Assessment (Appendix E)

<sup>&</sup>lt;sup>6</sup>Transesophogeal Echocardiogram (TEE) may be used if TTE is not available

<sup>&</sup>lt;sup>7</sup>For patients with abnormal findings related to valve integrity and position and patients with Adverse Events related to worsening valve function.

- Six Minute Walk Test (Appendix F)
- Kansas City Cardiomyopathy Questionnaire (KCCQ) (Appendix G)
- Clinical Laboratory Tests
  - o Blood count (hemoglobin, hematocrit, platelet count, white blood cells)
  - o PTT or PT/INR
  - o CK/CK-MB and/or Troponins
  - o Creatinine
  - o Liver Panel (ALT, AST)
  - o Albumin
- Non-invasive studies
  - o 12-Lead ECG
  - Chest x-ray

# **Procedure**

Transfemoral access technique will be used by the investigator in his/her normal practice of interventional cardiology and patient selection process.

#### Recommended Antiplatelet/Anticoagulation Regimen

Table 4 outlines the recommended antiplatelet regimen. The categories were developed by The PARTNER II Trial Patient and Procedure Management Steering Committee. There are no current validated guidelines in this specific study population, however, the literature was surveyed and used as guidance for the following proposed guidelines. It is expected that specific agents and dosing regimens may vary from site to site. Patients will be assessed by the heart team for Category of Stroke Risk prior to prescribing treatment regimen. The Category and specific treatment regimen will be documented in the discharge case report form. Committee Categories are based on CHADS 2 score for stroke risk [27].

NOTE: The CHADS 2 score only applies to patients in atrial fibrillation (AF) and has not been validated in non-AF patient populations; therefore the CHADS 2 score reference was used as one among many guidelines to establish the risk stratification for intensity of anticoagulation regimen.

Table 3. Summary of Recommended Antiplatelet/Anticoagulation Therapy

| Pre procedure | Aspirin 75-100 mg once daily |
|---|---|
| | <ul> <li>Patients with bare metal stent (BMS) within one month or drug eluting stent (DES) within 12 months should be continued on Clopidogrel/Prasugrel prior to their procedure</li> <li>Patients in atrial fibrillation on warfarin should be bridged with LMW or UF heparin prior to the procedure</li> <li>Patients with persistent or paroxysmal atrial fibrillation, not on anticoagulation, will not be required to have a TEE to rule out LA thrombus prior to procedure. If intraprocedural TEE during TAVI reveals thrombus, procedure will be aborted and delayed until patient has been on</li> </ul> |

| Tatus nus sadana | warfarin or dabigatran for 30 days. • In patients under concomitant TAVI/PCI, Clopidogrel loading with either 300mg or 600mg prior to the procedure is recommended in addition to ASA: Hanning will be given to a selving of projection ACTS 250 and |
|---|---|
| Intra procedure | Heparin will be given to achieve/ maintain ACT \subsection 250 sec. |
| Post procedure Category I for Stroke Risk No atrial fibrillation, No recent stents | <ul> <li>ASA 75mg once daily</li> <li>Clopidogrel 300mg load within 6 hours of procedure (either pre or post)</li> <li>Clopidogrel 75mg once daily for at least one month post procedure</li> </ul> |
| Category II for Stroke Risk No atrial fibrillation, recent stents | <ul> <li>ASA 75mg once daily</li> <li>Clopidogrel 75mg once daily should be continued prior to<br/>the procedure and after the procedure without interruption<br/>for at least one month after BMS and 12 months after DES</li> </ul> |
| Category III for Stroke Risk Atrial fibrillation, no recent stents | <ul> <li>ASA 75mg once daily</li> <li>Patients should be started on warfarin or dabigatran 24 hours post TAVI if clinically safe and this should be continued for at least one month or indefinitely if possible. If clinically safe, patients started on warfarin should be bridged with unfractionated or low molecular weight heparin until INR therapeutic.</li> <li>If patients are not a candidate for warfarin or dabigatran.</li> </ul> |
| Category IV for Stroke Risk Atrial fibrillation, recent stents | <ul> <li>If patients are not a candidate for warfarin or dabigatran, Clopidogrel 75mg once daily can be considered as an alternative</li> <li>ASA 75mg once daily</li> <li>Clopidogrel 75mg once daily for at least one month post BMS or 12 months post DES</li> <li>Patients should be started on warfarin or dabigatran 24 hours post TAVI if clinically safe and continued indefinitely. If clinically safe, patient's being started on warfarin should be bridged with UF or LMW heparin until</li> </ul> |

Note: Any changes to anticoagulation regimen from study visit to study visit will be noted on the CRF including reason for change.

# **Antibiotic Prophylaxis**

Study subjects should be treated prophylactically with antibiotics for endocarditis per the recommendations of the American Heart Association [28].

Version 1.0, 2017 June 22 Edwards Confidential Page 19 of 37

#### **Procedure Assessments**

Procedural information, findings, results, and SAPIEN 3 delivery system and device identification will be recorded on the Case Report Form and are listed below:

- Duration of the procedure, defined as the time from skin incision to access closure;
- All cardiac medications and all medications given for cardiovascular effect;
- A supra-aortic angiogram or TEE to assess valve performance and coronary patency
- Fluoroscopic imaging of implanted valve to assess acute deployment (e.g. proper annular placement, fully vs. under deployed, circularity/ovality)
- Contrast media quantity
- Total fluoroscopy time and dose
- Adverse Events

Subjects will be continuously monitored clinically, hemodynamically, and electrocardiographically during the index procedure for all local and systemic side-effects.

It is recommended subjects are monitored in the operating room for at least 15 minutes after completion of the procedure, with special attention to hemodynamic condition and cardiac rhythm. The sheaths may be removed when ACTs reach <150 sec after implantation of the study valve (for non-surgical closures).

#### Post-Procedure

Post-procedure clinical evaluations should be performed within 48 hours of the index procedure. Specific assessments include the following:

- Current cardiac medications and all medications given for cardiovascular effect
- Adverse events
- Neurological assessment
  - o NIHSS
  - o mRS
- Clinical Laboratory Test
  - o Blood count (hemoglobin, hematocrit, platelet count, white blood cells)
  - o PTT or PT/INR
  - o CK/CK-MB and/or Troponins
  - Creatinine
  - 12-Lead ECG

#### Discharge Visit

The following data will be collected for all study patients before discharge from the index hospitalization. If patient is discharged over a weekend, the discharge tests may be completed on the last weekday prior to discharge. For patients that are discharged within the 48 hours of exiting the cath lab / operating room, it is not required to repeat tests collected during the Post Procedure period that are also required for the Discharge visit.

- Pertinent physical examination [include blood pressure, weight and all major systems findings]
- Current cardiac medications and all medications given for cardiovascular effect
- NYHA functional classification
- CSS Angina Classification
- Adverse events
- Neurological assessments
  - o NIHSS
  - o mRS
- Clinical Laboratory Test
  - o Blood count (hemoglobin, hematocrit, platelet count, white blood cells)
  - o PTT or PT/INR
  - o Creatinine
- 12-Lead ECG
- Comprehensive TTE. If not adequate, a TEE will be performed

#### Follow-Up Visits

The determination of the study endpoints will require rigorous clinical follow-up and quality data collection. The Investigator or delegated study personnel will ensure the patient is scheduled for follow-up visits according to Table 5.

Table 4. Follow-up Visit Windows

| Follow-Up Visit | Visit Window (days following Procedure) |
|-----------------|-----------------------------------------|
| 30 Day | 30 days, +14 days |
| 6 Month | 180 days +/-30 days |
| 1 Year | 365 days +/-60 days |
| 2 Year | 730 days +/-60 days |
| 3 Year | 1095 days +/-60 days |
| 4 Year | 1460 days +/-60 days |
| 5 Year | 1825 days +/-60 days |

The importance of attending the 30 Day follow-up visit should be discussed with the patient. Planned absences should be recorded to facilitate continued ability to contact a study patient during the course of the study. If a patient cannot be reached for a follow-up visit, the investigator will document on the follow-up data form, the efforts undertaken to contact the patient, referring physicians, including internists as well as cardiologists, family members, or other alternate contacts noted in the study patient's records. These efforts should include 3 attempts of telephone contacts at separate dates and times, and a registered letter. If a patient can no longer be located, the investigator must contact an intermediary (e.g. patient's private physician) without delay.

Patients for whom the study procedure was begun but do not receive and retain the study valve will be followed up until the 30-day assessment or resolution of any AE for safety purposes. Patients with an ongoing AE at the 30 Day visit should have AEs reassessed at 30 day window closure (day 44). These patients should then be exited from the study. In the event that the patient's implanted

valve is explanted, the patient needs to be followed up until resolution of any AE for safety purposes. These patients should then be exited from the study.

### 30-Day Visit

All patients will undergo the following assessments within the 30-Day follow-up period +14 days):

- Pertinent physical examination [include blood pressure, weight and all major systems findings]
- Adverse events
- Current cardiac medications and all medications given for cardiovascular effect
- NYHA functional classification
- CSS Angina Classification
- Neurological assessments
  - o NIHSS
  - $\circ$  mRS
- 6 Minute Walk Test (6MWT)
- KCCO
- Clinical Laboratory Test
  - o Blood count (hemoglobin, hematocrit, platelet count, white blood cells)
  - o Creatinine
  - o CK/CK-MB and/or troponins
  - o Albumin
- 12-Lead ECG
- Comprehensive TTE. If not adequate, a TEE will be performed

For patients with abnormal findings related to valve integrity and position and patients with adverse events related to worsening valve function, fluoroscopic imaging of the implanted valve will be completed.

#### 6 Month Visit

All patients will undergo the following assessments within the 6 Month follow-up period:

- Adverse events
- Current cardiac medications and all medications given for cardiovascular effect

The 6 month visit may be completed via a telephone conversation with a delegated study team member. The telephone call must be documented in the patient's study records.

#### 1 Year Visit

All patients will undergo the following assessments within the 12 Month follow-up period:

- Pertinent physical examination [include blood pressure, weight and all major systems findings]
- Adverse events

- Current cardiac medications and all medications given for cardiovascular effect
- NYHA functional classification
- CSS Angina Classification
- 12-Lead ECG
- Comprehensive TTE. If not adequate, a TEE will be performed

For patients with abnormal findings related to valve integrity and position and patients with adverse events related to worsening valve function, fluoroscopic imaging of the implanted valve will be completed.

# 2-5 Year Annual Follow-up Visit

All patients will undergo the following assessments within the 2-5 Year annual follow-up period:

- Pertinent physical examination [include blood pressure, weight and all major systems findings]
- Adverse events
- Current cardiac medications and all medications given for cardiovascular effect
- NYHA functional classification
- CSS Angina Classification
- Comprehensive TTE. If not adequate, a TEE will be performed

For patients with abnormal findings related to valve integrity and position and patients with adverse events related to worsening valve function, fluoroscopic imaging of the implanted valve will be completed.

#### Missed Visits

Every patient should be encouraged to remain in the study until they have completed the protocol-required follow-up period. If the patient discontinues prematurely from the study, the reason for discontinuation must be documented on the appropriate case report form (CRF). Possible reasons for premature discontinuation may include, but are not limited to the following:

- Withdrawal of consent: Patient decides to withdraw from the study. If a subject withdraws from the clinical investigation, the reason(s) should be recorded. If such withdrawal is due to problems related to the investigational device safety or performance, the investigator shall ask for the subject's permission to follow his/her status/condition outside the investigation.
- Lost to follow-up: All patients should be encouraged to return to the clinic for evaluation during follow-up (excluding 6 Month telephone visit). If a patient is unable to return to the clinic, 3 separate telephone calls should be made to attempt to bring the patient back into the clinic or obtain safety information. All attempts should be documented in the source documents. If the patient does not respond to the 3 telephone calls then the Investigator should send a certified letter to the subject.

#### Standard of Care

All enrolled patients will receive the standard of care during the clinical trial as well as following

the conclusion of their participation. Any patients with symptoms of valve failure at any time throughout the study duration should undergo standard diagnostic imaging (e.g. (TTE)) to assess valve function. Each patient will be provided with an implant card. This implant card can be carried by the patient to be shown to any clinician to inform a treating physician of the implanted SAPIEN 3 THV. Subjects that are enrolled, but not treated with the SAPIEN 3 THV will likely be screened for alternative treatments (when available) or continue with the care they have been receiving to date.

#### 7.1.6 Safety and Effectiveness evaluation methods

#### **Primary Endpoint**

The primary endpoint is all-cause mortality at 30 days post-index procedure.

#### Secondary Endpoints

#### Safety Endpoints

- Cardiovascular and non-cardiovascular mortality at 72 hours (peri-procedural) and 30 days
- Stroke at 30 days
- TIA at 30 days
- All-cause mortality & disabling stroke at 30 days
- Vascular complications (major) at 30 days
- Bleeding complications (life threatening or disabling, and major) at 30 days
- Myocardial infarction at 30 days
- Acute kidney injury at 30 days (stages II and III)
- Coronary obstruction requiring intervention at 30 days
- Arrhythmia and conduction disturbance at 30 days
- Permanent pacemaker implantation at 30 days
- Valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVR) at 30 days
- Mitral valve apparatus damage or dysfunction at 30 days
- Unplanned use of cardiopulmonary bypass (CPB) during TAVI implant procedure
- Pericardial tamponade at 30 days
- Endocarditis at 30 days
- Valve thrombosis at 30 days
- Valve malposition (migration, embolization, and ectopic deployment) at 30 days
- Ventricular septal perforation at 30 days

# Device and Procedure Success Composite

- Absence of procedural mortality AND
- Correct positioning of a single prosthetic heart valve into the proper anatomic location AND
- Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20mmHg or peak velocity <3m/s, AND no moderate or severe prosthetic valve regurgitation) at 30 Days

# Efficacy

- New York Heart Association (NYHA) Classification at 30 days
- Hemodynamic valve performance evaluation by echocardiography for aortic valve stenosis and aortic valve regurgitation (paravalvular & central) at 30 Days as determined by Echo core lab

# Quality of Life

- KCCQ at 30 days
- 7.2 Test process
- 7.2.1 Test flowchart

Figure 2. Trial Process Diagram



# 7.2.2 Specification for use of devices

Version 1.0, 2017 June 22 Edwards Confidential Page 25 of 37

# Study Device

The SAPIEN 3 and its delivery components will have a unique product identifier. This information will be recorded in the study subject's medical file. The Instructions for Use for the SAPIEN 3 THV System are provided with the device.

# Storage & Labeling

The SAPIEN 3 THV System is to be stored as specified on the unit labels. All investigational stock will be stored in a secure and controlled area.

# **Device Accountability**

The Investigator shall maintain accurate records of the receipt and disposition of the investigational devices. A device disposition log supplied by Edwards will be used to record device receipt, uses, discards, or returns. Device disposition will be verified by the Sponsor periodically throughout the study. All unused devices shall return to Edwards, along with the completed device disposition log at completion of the enrolment period. The Investigator's copy of the device disposition log must document the devices used in study subjects as well as unused devices that are returned to Edwards. Use of the SAPIEN 3 THV System is prohibited outside of this protocol.

#### 7.3 Monitoring Plan

Edwards Lifesciences will contract with a Contract Research Organization (CRO) to provide a Clinical Research Associate(s) (CRA) to monitor the study sites to ensure that all investigators are in compliance with the protocol and the Investigator's Agreement, and that all study subjects have been properly consented with the current version of the informed consent document. Edwards Lifesciences will evaluate circumstances where an investigator deviates from the clinical protocol and will retain the right to remove either the investigator or the investigational site from the study.

Routine on-site monitoring visits shall include verification of the following:

- Compliance with the protocol, any subsequent amendment(s), GCP and maintenance of regulatory and EC requirements. Deviations shall be discussed with the Investigator(s) or delegated personnel, documented and reported
- Only authorized and delegated individuals are participating in the study
- The SAPIEN 3 THV System is being used according to the protocol and IFU
- Study Site resources, equipment and study personnel, remain adequate throughout the duration of the study
- Patient Informed Consent is completed in accordance to the protocol and regulations
- Only Patient Informed Consents Forms approved by the EC are used appropriately
- Source documents and other clinical records are accurate, complete up to date, stored and maintained properly
- CRFs and queries are complete, recorded in a timely manner, and consistent with source documents
- All adverse events and device deficiencies are reported to Edwards without unjustified delay
- All serious adverse events and deviations are reported to the EC, if required

- All other required reports, notifications, applications, submissions and correspondence are maintained in the investigator's files and are accurate, complete, timely, legible, dated and identify the clinical investigation
- Current laboratory normal values, laboratory certifications, accreditations, or other validations are present in the investigator's file
- Subject withdrawal has been documented; the monitor shall discuss this with the principal investigator or his/her authorized designee
- Subject non-compliance with the requirements stated in the informed consent has been documented; the monitor shall discuss this with the principal investigator or his/her authorized designee
- Suitability of the attempts to contact lost to follow-up patients and any intermediaries
- The principal investigator and investigation site team are informed and knowledgeable of all relevant document updates concerning the clinical investigation
- Any corrective and preventive actions, as needed, have been implemented and are effective. Monitors shall be appropriately qualified per the following requirements:
  - Qualified in the field of the applicable regulations and GCP through training and experience as well as scientific or clinical knowledge;
  - Knowledgeable on the use of the investigational device(s) and relevant requirements, protocol and informed consent process;
  - All monitoring activities shall be documented in a written report. The frequency of monitoring visits will depend on enrollment and center compliance, but each center will at least be visited once per year. Further details are laid out in the monitoring plan.

Edwards Lifesciences will review significant new information, including unanticipated adverse events and ensure that such information is provided to the study investigators and to all reviewing ECs and regulatory agencies as necessary. Efforts will be made to ensure that data collection compliance is monitored and communicated to the Investigators in a timely manner throughout the trial.

#### 8. Statistical considerations

# 8.1 Statistical design, method, and analysis procedures

The clinical study is a single-arm prospective study intended to demonstrate the safety and performance of the SAPIEN 3 THV in the Chinese population.

#### 8.2 Sample Size

The sample size of 50-60 patients is determined per Chinese regulatory requirements and agreement for a regional study of a medical device already approved in other regions based on a well-designed prospective study.

8.2.1.1 Minimum and maximum number of subjects for each clinical trial institution and reasons

To ensure that a minimum of 50 patients are implanted with the SAPIEN 3 THV and complete the 30 Day follow-up for Primary Endpoint, up to 60 patients will be enrolled and implanted with

SAPIEN 3 THV. Each site may not contribute more than 25 implanted patients to the study population.

### 8.3 Expected expulsion rate

The Chinese regulatory requirements determine 50 patients should meet the primary endpoint. If a minimum of 50 patients complete 30 Day visit and upto 60 patients have the procedure, the expected drop-out rate is <17%.

8.4 Statistical method for all data, together with deficient, unused or fault data (including drop out and withdrawal) and method for treating unreasonable data

The primary and secondary endpoints will be reported based on the AT Population. Descriptive and summary statistical analysis will be performed on all endpoints. Patient listings for adverse events, deaths, and reinterventions will include all enrolled patients.

All clinically relevant baseline and follow-up variables will be tabulated. Descriptive statistics for continuous variables include mean, standard deviation, sample size, median, minimum, and maximum) and frequency tables or proportions for discrete variables.

Kaplan Meier estimates will be performed at the pre-specified follow-up times to project the estimates for time-related endpoints such as the 30-day mortality rate, the primary endpoint; the standard error and confidence limits will be computed using Greenwood's algorithm. Based on 50 patients as point estimate and length of estimate on the primary endpoint, the 30 days death rate and 95% confidence interval will be summarized.

Echocardiographic data will be analyzed by an Echo core laboratory with respect to the degree of total aortic valve regurgitation (TVR) and paravalvular aortic valve regurgitation (PAR) according to the VARC-2 definitions [29].

These data and other categorical data (e.g., NYHA class) will also be presented as shift from baseline for each of the pre-specified follow-up periods.

8.5 Procedures for reporting deviation from the original statistical plan

More detailed information regarding the statistical methods and analysis will be presented in the Statistical Analysis Plan (SAP). Statistical method changes and/or deviation from the original statistical analyses plan will be documented in the section of amendment of the versioned SAP which requires re-approval before the performance of analyses and to be included in the final study report.

8.6 Criteria and reasons for selection of subjects incorporated into analysis

All patients documented as part of the roll-in patient strategy will not be included in analysis population and will be evaluated separately.

**Analysis Sets** 

• As Treated (AT) Population: all patients that were enrolled in the trial for whom the SAPIEN 3 valve implant procedure was begun, defined as the time in which the first Edwards' investigational device is inserted into the patient.

• *Valve Implant (VI) Population:* all AT patient who received and retained the SAPIEN 3 valve upon leaving the procedure room

#### 9. Data Management

#### 9.1 Data Collection

Data will be captured and managed through an electronic data capture (EDC) system. Passwords will be issued to appropriate data management personnel to ensure confidentiality and protection of the data by allowing variable levels of access to the computer system.

Electronic CRFs (eCRFs) will be used to collect all patient data during the trial. eCRFs must be fully completed for each patient, and signed electronically by the investigator and/or designee.

The investigator, or an individual designated by him/her, is responsible for recording all data from the trial onto the eCRFs on a dedicated website. The investigator is required to provide an electronic signature on the appropriate eCRF pages to verify that he/she has reviewed the recorded data.

Completed eCRFs will be reviewed at the investigational site and remotely by authorized Edwards Lifesciences personnel at regular intervals throughout the trial. All eCRFs will be tracked at Edwards Lifesciences and missing or unclear data will be requested as necessary throughout the trial.

# 9.2 Missing Data

All possible steps will be taken to minimize missing data in the study, including monitoring of data forms for completeness and efforts to track and maintain contact with study subjects during the follow-up period.

#### 10. Feasibility Analysis

#### 10.1 Successful possibility analysis

Product handling and procedure guidance are provided in the Training Materials and IFU and will be used for device training to minimize risks associated with device use.

Additionally, efforts will be made to minimize these possible risks though site/investigator selection and management. First, site and investigator selection criteria are established to ensure that the study personnel and their institutions are qualified to screen, perform and manage the study procedures as well as support the associated requirements for research.

Second, the trial management structure is designed to provide disciplined oversight of the trial activities including close monitoring of site and personnel performance and also support opportunities for investigators and study personnel to share best practices through investigator meetings, ongoing education and case reviews.

Site and investigator criteria include the following:

- Interventional cardiologists must be experienced and skilled in percutaneous balloon valvuloplasty.
- Strong interdepartmental collaboration between cardiac surgery and interventional cardiology operators will be assessed by an experienced trial study team. The study site

team must be trained in the use of the investigational devices prior to enrollment of study patients.

- The procedure setting must include a fixed C-arm angiography and PCI imaging capability in the catheterization lab or operative suite and/or a hybrid catheterization/operating room suite.
- The study site must have an operating room.

The study site must have an adequately staffed research department with a minimum of one dedicated study coordinator

# 10.2 Analysis of the possibility of failure

For the purposes of this study, adverse events that may be anticipated are associated with the use of the SAPIEN 3 THV System as well as the anesthesia and interventional procedures used to deliver and deploy the SAPIEN 3 THV.

Anticipated risks have been minimized to the furthest extent possible, but the nature of the procedure and the severity of the patient's disease state has inherent risks. Exposure to ionizing radiation associated with fluoroscopy, x-rays and CT is no more than is associated with routine clinical practice for transcatheter aortic heart valve replacement.

Risks are outlined in the SAPIEN 3 THV System Instructions for Use (IFU)

### 11. Quality control of clinical trials

Clinical sites will be chosen that have proper facilities in place to complete THV procedures. Additional training of appropriate clinical site personnel will be the responsibility of the Sponsor. To ensure proper device usage, uniform data collection, and protocol compliance, the Sponsor will present a formal training session to study site personnel which will review the instructions for use of the device, the Investigational Plan, techniques for the identification of eligible patients, instructions on in-hospital data collection, CT recommendations, echocardiography data collection for core laboratory analysis, methods for soliciting data from alternative sources, schedules for follow-up with the study site coordinators, and regulatory requirements. Detailed feedback regarding completion of forms will be provided by the Sponsor, and through regular site monitoring. Edwards Lifesciences reserves the right to enforce retraining for sites who have demonstrated study or procedure compliance issues.

#### 12. Ethical issues and informed consent for clinical trials

#### 12.1 Ethical considerations

The SAPIEN 3 THV System is not commercially available in China. The clinical investigation shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki (as updated in Fortaleza Brazil in 2013) and in compliance with China's Good Clinical Practice (GCP) for Medical Devices and any national regulations.

#### 12.2 Examination and approval of clinical trial protocol

The clinical investigation plan and Patient Informed Consent form used to study the SAPIEN 3 THV System must be reviewed and approved by the appropriate national authority and local or regional Ethics Committee (EC) where the clinical investigation is to be conducted before

enrolment of patients may begin. Any additional requirements imposed by the EC or regulatory authority shall be followed.

Changes to the investigational plan that may increase the risk or present new risks to the patient must be approved in writing by Edwards Lifesciences and the EC before the change is implemented.

#### 12.3 Informed consent process and text of informed consent

The Patient Informed Consent Form must be approved by Edwards Lifesciences and the site's EC.

The study investigator(s) and support staff will approach patients with symptomatic aortic stenosis to assess their interest in participating in the study. They will provide an overview of the study and device, including the background, benefits, risks, and study procedures. If patients are interested in participating in the study, then they will be provided with the full Patient Informed Consent Form document. Patients will be allowed to read the document in its entirety, and then delegated study personnel will answer all of their questions. If the patient is comfortable with proceeding, then they will be asked to sign and date the Patient Informed Consent Form. Informed consent must be obtained prior to the screening procedures or baseline tests that are specific to this study.

During the course of the study, if new information becomes available that can affect a patient's future health and medical care, then the information will be provided to the patient and the process documented. If relevant, all affected patients will be asked to confirm their continuing informed consent in writing.

All patients who sign a Patient Informed Consent Form should be entered in the database. Data should not be entered until a Patient Informed Consent Form is signed. Patients that are screened and do sign a Patient Informed Consent Form should be documented on the Screening Log.

#### 13. Provisions on adverse event and device defect report

#### 13.1 Adverse events

Adverse events may be volunteered by patients, elicited from questioning by Investigator or delegated study personnel, or collected via observation by the Investigator. In addition, patients will be instructed to contact the investigator, and/or study coordinator if any significant adverse events (e.g., expanded safety composite events) occur between study evaluation visits.

All adverse events are reported from the start of the procedure, which is defined as when anesthesia is first administered, and are reported until subject participation has ended (i.e. completion of the study or withdrawal of consent). Adverse events must be reviewed at every follow-up visit until resolution, AE has stabilized (according to Investigator), or the study has been completed. Should the adverse event be ongoing at time of study completion, the database should be updated to reflect status.

Reporting guidelines for adverse events:

 Record the number of units of blood needed for any transfusion associated with any overt bleeding event

- Failure of a percutaneous closure device shall be reported as an access site vascular closure device complication
- Vascular complications shall be designated as access or non-access related;

#### 13.2 Serious Adverse Events

All Serious Adverse Events (SAE) and Unanticipated Serious Adverse Device Effect (USADE) must be reported to Edwards Lifesciences within 24 hours of the Investigator or delegated study personnel becoming aware of the event or according to local regulations (whatever is most stringent). SAEs and USADEs will be reported to the EC and regulatory authorities as required by national regulations or by the EC itself.

Information may be entered into the Case Report Form or reported directly to the Edwards Lifesciences, with documentation of such notification being recorded and filed. Notifications and source documents will be provided to Safety Officer.

At the time of initial notification, the following minimal information should be provided:

- Identifiable patient: subject number
- Identifiable reporter: study site
- Adverse event summary
- Causal relationship to device and procedure
- Awareness date

The USADE Case Report Forms should be completed within five working days. All USADEs must be followed until resolution or until a stable clinical endpoint is reached. All required treatments and outcomes of the USADE must be recorded.

Edwards will notify all participating clinical Investigators, ECs, and regulatory bodies as necessary of all USADEs that occur during the study within the specified reporting time frame following event notification. Investigators are responsible for reviewing information received about USADEs.

#### 13.3 Reporting procedure and information of contact

# Source Documents

The site will provide to Edwards Lifesciences a copy of anonymized supporting documentation (such as hospital record, laboratory results, autopsy results) of all SAEs and safety related composite events.

#### **Investigator Assessment Responsibilities**

The Investigator will determine if an adverse event is serious and not related, possibly related, or related to the device or procedure.

Pre-existing medical conditions or symptoms reported prior enrolment will be recorded in medical history form and will not be recorded as an adverse event. In the event there is a worsening in the pre-existing medical condition or symptoms after enrolment, then an adverse event will be recorded.

#### Sponsor Assessment Responsibilities

All adverse events will be reviewed by the Study Safety Officer who will determine if the adverse event is serious; anticipated or unanticipated; and not related, possibly related, or related to the device or procedure.

# Medical Reviewer Responsibilities

All endpoint related adverse events will be reviewed by a Medical Reviewer who will determine if the adverse event is serious; and not related, possibly related, or related to the device or procedure.

# 1.1. Device Deficiency

Device deficiency is an inadequacy of a medical device with respect to its integrity, quality, durability, reliability, safety or performance. It includes malfunctions, user errors and inadequate labeling.

Device deficiencies include those deficiencies that did not lead to an adverse event but could have led to a medical occurrence:

- a. If intervention had not been made, or
- b. If circumstances had been less fortunate.

Reporting conventions for device deficiencies that could result in a Serious Adverse Event (SAE) are the same as those for an actual SAE.

#### Device Deficiency and Vigilance Reporting

Device deficiencies which could have led to a serious adverse device effect should undergo the same reporting as serious adverse events. They should be reported to Edwards Lifesciences within 24 hours of awareness and to the EC and regulatory authorities as required by regulations or the EC.

Adverse device effects, device malfunctions and device failures must be reported to Edwards Lifesciences in accordance with the regulations and Edwards Lifesciences policies.

The Edwards Lifesciences 'Complaint Reporting Process' form is available in the site study document file.

#### 14. Provisions on deviation from clinical trial protocol and correction of clinical trial protocol

The investigator will not deviate from the protocol without the prior written approval of Edwards Lifesciences except in medical emergencies or in unforeseen, isolated instances where minor changes are made that will not increase the patient's risk or affect the validity of the trial. In medical emergencies, prior approval for protocol deviations will not be required, but the Edwards Lifesciences clinical research personnel must be notified within 24 hours of the incident.

All protocol deviations need to be recorded in the respective section of the eCRF and reported according national and ethics committee requirements. Periodic monitoring of protocol compliance will be performed for each site. The sponsor maintains the right to place a moratorium on enrollment in sites deemed to have excessive protocol compliance issues. A major protocol violation is the instance where a deviation significantly affects the integrity of the study and guidelines for Good Clinical Practice, such as when there is failure to obtain informed consent or violation of inclusion/exclusion criteria. In cases of major protocol violation, the principal investigator is required to make a written statement attesting to retraining or other action(s) to be

taken at his/her site to avoid such violations in the future.

#### 15. Direct access to source data and files

#### Records

All records related to the study and qualifications of site personnel must be kept on file and available for review. These documents may include but are not limited to:

- Clinical trial investigational plan and all amendments, all approved versions
- Signed clinical trial agreement
- EC approval letter, including final informed consent
- EC membership list
- Correspondence relating to the trial
- CVs for all investigators and research coordinator
- Site personnel signature list
- Clinical monitor sign-in log
- Patient screening/enrollment log
- Lab certification and lab test normal ranges
- Reports (includes reports from investigator and sponsor)

All records related to the patients' consent and study data must be maintained for each patient enrolled in the trial. These records include and are not limited to:

- Signed Patient Informed Consent Form (latest approved site version)
- All completed eCRFs
- Supporting documentation of any complications and/or safety events.

Edwards Lifesciences requests that the investigator retain copies of procedure reports, procedure nursing notes and the results of any interventional procedures that occurs post trial procedure. Edwards Lifesciences reserves the right to secure data clarification and additional medical documentation on patients enrolled in this trial.

# Record Retention Policy

All clinical sites will maintain study records for a minimum of 15 years after marketing approval is obtained. After 15 years, clinical sites should follow hospital and regulatory guidelines for record retention. Record retention dates will be provided to all parties concerned by Edwards Lifesciences.

#### 16. Finance and insurance

#### Clinical Trial Funding

As the Sponsor, Edwards Lifesciences will fund the trial for its duration.

# Clinical Trial Insurance

As required by local/country regulation, Edwards Lifesciences will obtain clinical trial insurance for the duration of the clinical trial and provide evidence of coverage.

#### 17. Contents to be covered by clinical trial reports

The template of the Clinical Trial Report can be found in Appendix G.

# 18. Principle of medical confidentiality

All information and data sent to the data management center concerning patients or their participation in this trial will be considered confidential. Only authorized data management center personnel will have access to these confidential files. Authorized personnel from Edwards Lifesciences and its contractors and regulatory authorities have the right to inspect and copy all records pertinent to this trial. All data used in the analysis and reporting of this evaluation will be without identifiable reference to the patient.

#### 19. Provisions on publication of clinical trial results

Clinical sites have the right, consistent with academic standards, to publish their individual registry results provided such publication does not constitute a violation of the Study Agreement. The site agrees to submit any proposed submission for publication to Edwards Lifesciences for review and approval before any submission. Consent cannot be denied without a sensible reason.

The results of the clinical investigation will be submitted, whether positive or negative for publication. The publication policy will be part of Study Agreement.

# 20. Responsibilities of all parties

# **General Study Organization**

Edwards Lifesciences is the Study Sponsor, and has the overall responsibility for the conduct of the study, including assurance that the study meets the regulatory requirements of the appropriate regulatory bodies. Edwards Lifesciences will have certain direct responsibilities and will coordinate other responsibilities to the specified committees, Echo core lab and other support services as necessary

Edwards Lifesciences will be responsible for submitting the Clinical Investigation Plan and all changes to it to the regulatory body and local EC to obtain ongoing approvals as needed.

Edwards Lifesciences will submit all reports required by the appropriate regulatory authorities as identified in this section of the regulation. This may include unanticipated and serious adverse device effects, withdrawal of EC approval, current investigators list, annual progress reports, recall information, final reports and protocol violations.

Edwards Lifesciences and Core Laboratories will maintain copies of correspondence, data, shipment of devices, adverse device effects and other records related to the study as appropriate.

#### Medical Reviewers

Medical Reviewers will review and classify adverse events in accordance with the study protocol.

# **Echocardiography Core Laboratory**

A Core laboratory will be established for Echocardiography endpoint analysis. Standardized protocols for acquiring and transmitting electronic records will be developed and documented prior to study initiation.

Clinical Sites will upload a qualifying echocardiography prior to the enrolment of the first subject in accordance with the standardized protocol.

Edwards Lifesciences will review echocardiography data for the duration of the study.

# Clinical Sites

Edwards Lifesciences will select qualified investigators, ship devices only to participating investigators, obtain a signed Clinical Study Agreement and provide the investigators with the information and training necessary to conduct the study. Edwards Lifesciences will retain copies of all study-related correspondence with study sites.

#### 21. Statement of Investigator

I hereby agree:

- 1. Carry out this clinical trial strictly according to the requirements of the Declaration of Helsinki, current laws and regulations of China, and the protocol.
- 2. Accurately record all data required into the case report form (CRF) and accomplish clinical trial report on time.
- 3. The medical device for test is only used for this clinical trial. Completely and accurately record the receiving and the use of the medical device for the test during the clinical trial and maintain the record.
- 4. Allow the sponsor to authorize or dispatch supervisor, inspector and supervisory department to conduct supervision, inspection, and check on the clinical trial.
- 5. Strictly perform the clinical trial contract/agreement signed by all parties.

I have carefully read the clinical trial protocol including above statement and I agree with all contents above.

| Opinions of sponsor |
|-------------------------------------------------------|
| Signature (seal) |
| Date: |
| Opinions of investigator |
| Signature |
| Date: |
| Opinions of medical device clinical trial institution |
| Signature (seal) |
| Date: |